CLINICAL TRIAL: NCT00368303
Title: A Multicentre, Double-blind, Active Controlled Trial to Evaluate the Clinical Effects of Immediate Release Paroxetine and Controlled Release Paroxetine in the Treatment of Major Depression
Brief Title: A Local Register Study For Major Depression Of Paroxetine Controlled Release
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCR103124
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Depressive Disorder, Major; Major Depressive Disorder (MDD)
Keywords: Major Depression; paroxetine controlled release (CR); paroxetine immediate release (IR)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paroxetine CR
Drug: Paroxetine IR
  Other Names: Paroxetine CR

SUMMARY:
The study is to investigate the non-inferior efficacy of Paroxetine Controlled Release to Paroxetine Immediate Release, as well as the drug tolerability profile when treated on patients with Major Depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Major Depressive Disorder,score on depression rating scale reach a specific point(17 item Hamilton Depression Scale>18).

Exclusion criteria:

* patients use monoamine oxidase inhibitors (MAOIs), benzodiazepines, Chinese herbal medicines, acupuncture, moxibustion or other psychoactive medications other than zolpidem, zopiclone;diagnosed with other Axis I disorder other; not responsive to paroxetine therapy before; pregnant or lactating, have serious medical disorder or condition that would preclude the administration of paroxetine; have a history of seizure disorders (except for febrile seizures in childhood); require treatment with warfarin anticoagulants, phenytoin, cimetidine, sumatriptan, type 1C antiarrhythmics, quinidine or sulfonylurea derivatives; are substance abuse or dependence (alcohol or drugs) within 6 months prior to this trial; have had electroconvulsive therapy within 2 months of entry into the study; pose a current, serious suicidal or homicidal risk; have taken other psychotropic drugs or antidepressants other than MAO inhibitors within 7 days of baseline and MAO inhibitors within 14 days of baseline; have taken any investigational drug, or participated in a clinical trial within the past 3 months; are hypersensitivity to paroxetine; have undergoing formal psychotherapy/psychoanalysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362
Dates: Start 2006-12

PRIMARY OUTCOMES:
Scores on depression rating scale at treatment week 1,2,3,4,6 and 8.

SECONDARY OUTCOMES:
Scores on clinical impression severity and improvement items at treatment week 1, 2,3,4,6,8

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- China (8):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Baoding, Hebei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Beijing